CLINICAL TRIAL: NCT01943656
Title: A Longitudinal Clinical Feasibility Study to Evaluate the Psychological and Functional Effects of Using the Tobii™ Eyegaze System by Inpatients With Tetraplegia
Brief Title: Eyegaze Systems for Spinal Cord Injury: A Feasibility Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13/EE/0049 (UK NRES)
Record Dates: First submitted 2013-07-22; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tobii™ Eyegaze System (Experimental): Single arm, open label study.
  Interventions: Device: Tobii™ Eyegaze System

INTERVENTIONS:
Device: Tobii™ Eyegaze System — Volunteers will be instructed and trained to use the Tobii™ Eyegaze System. The number of sessions required to successfully master the device depends on the learning curve of the patient. The progress will be documented accordingly. After successful completion of the training and supervised use, the inpatients will be offered the Tobii™ Eyegaze System for unsupervised use, 4 hours a week, for the following 2 months.
  Other Names: Eyegaze System, Eye-tracking Operation System

SUMMARY:
As technologies are advancing quickly in the healthcare setting, new solutions have become available helping disable people to enhance their ability to communicate. One of these advances is the introduction of the 'eye gaze system'. Through processing eye movements, this device allows a person to write, speak, use the Internet and even control systems in the home or office. In the currently proposed study we aim to evaluate the psychological and functional effects of using the Tobii™ Eyegaze System by inpatients with tetraplegia who are unable to use arms and legs and sometimes are not able to talk because of an impaired respiratory function.

Volunteering inpatients will be recruited at the National Spinal Injuries Centre. Volunteers will be instructed and trained to use the Tobii™ Eyegaze System. The number of sessions required to successfully master the device depends on the learning curve of the patient. The progress will be documented accordingly. After successful completion of the training and supervised use, the inpatients will be offered the Tobii™ Eyegaze System for unsupervised use, 4 hours a week, for the following 2 months. It is hypothesised that using the Tobii™ Eyegaze System by inpatients with tetraplegia results in improved disability perception and independence scores. For the current feasibility study 12 participants will be recruited and assessed for 'Appraisal of Disability', 'Mood', 'Assistive Technology perception' and 'eyeskills' to instruct the computer system. Positive study outcomes will encourage future studies of the role of the Tobii™ Eyegaze System in both a rehabilitation and home environment.

DETAILED DESCRIPTION:
Volunteering inpatients will be recruited at the National Spinal Injuries Centre. Volunteers will be instructed and trained to use the Tobii™ Eyegaze System. The number of sessions required to successfully master the device depends on the learning curve of the patient. The progress will be documented accordingly. After successful completion of the training and supervised use, the inpatients will be offered the Tobii™ Eyegaze System for unsupervised use, 4 hours a week, for the following 2 months. It is hypothesised that using the Tobii™ Eyegaze System by inpatients with tetraplegia results in improved disability perception and independence scores. For the current feasibility study 12 participants will be recruited and assessed for 'Appraisal of Disability', 'Mood', 'Assistive Technology perception' and 'eyeskills' to instruct the computer system. Positive study outcomes will encourage future studies of the role of the Tobii™ Eyegaze System in both a rehabilitation and home environment.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury at C7 level or above
* American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade A, B, C or D
* Age equal or higher than 16 years old
* Expected to stay least 10 weeks at the National Spinal Injuries Centre

Exclusion Criteria:

* History of severe neurological injuries other than Spinal Cord Injury (eg. Multiple Sclerosis, Cerebral Palsy, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Stroke)
* Planned discharge within 10 weeks time
* Psychiatric or cognitive conditions that may interfere with the study
* Patients incapable of providing informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Appraisals of Disability: Primary and Secondary Scale (ADAPSS) Questionnaire | 8 weeks
  Change in score between 0 and 8 weeks.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  Change in score between 0 and 8 weeks.

OTHER OUTCOMES:
Assistive Technology Device Predisposition Assessment© (ATDPA) Questionnaire | 8 weeks
  Change in score between 0 and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joost J. van Middendorp, MD, PhD, Principal Investigator — Stoke Mandeville Spinal Foundation
Locations (1):
- National Spinal Injuries Centre, Stoke Mandeville Hospital, Aylesbury, Buckinghamshire, United Kingdom

REFERENCES:
- See also: Website directing to project description and updates — http://www.smsf.org.uk/research%20projects.htm